CLINICAL TRIAL: NCT02104973
Title: Design and Evaluation of a Strategy to Prevent Overweight and Obesity in Schoolchildren in Mexico City
Brief Title: Obesity Prevention in Schoolchildren
Acronym: CRECES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Secretaria de Salud, Mexico (Other Government); Secretaría de Educación Pública, México (Other Government); Universidad Iberoamericana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-785-060; 2007-01-68854 (Other Grant/Funding Number: CONACYT)
Record Dates: First submitted 2014-01-23; First posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): After obtaining the approval of schools and parents, will be established in schools, units in which individual attention is given to children, parents and teachers that request: the advice is aimed at training users on healthy diet and constant physical activity. Workshops with children, in which selected topics will be discussed based on the analysis of depth interviews with children, parents and teachers, and information on habits and resources gathered through questionnaires will be conducted. The intervention included the provision of information and feedback with the population through a website. The work will include participation in the selection of foods sold in schools.
  Interventions: Behavioral: Lifestyle counseling
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Lifestyle counseling — We will intent to modify the diet of the children. The intervention is designed to promote the increase the intake of fruits and vegetables and to reduce the high density foods consumption.
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to design, implement and evaluate an intervention oriented to change alimentary practices and patterns of physical activity of children through educative activities with parents, teachers and children in school of Mexico city.

DETAILED DESCRIPTION:
In Mexico, obesity is becoming the most public health problem. The increase in body mass is associated with the changes in the alimentary environment, resources for physical activity in a context of poor health literacy of the population and low efficacy of the health system. Schools, as social settings, are a opportunity for obesity prevention.

The study includes three phases: 1) evaluation of training, in which the psychological context in which obesity is generated is evaluated. The evaluation will be performed by collection of qualitative and quantitative information, 2) design a strategy from the information obtained. The intervention will include working sessions with teachers, parents and children, establishment of schools in window counseling in nutrition and physical activity and the secretion of a website to not communicate with the public and Provide information, 3) evaluation of the strategy in a community trial with two groups of schools, one intervention and one control.

ELIGIBILITY:
Inclusion Criteria:

* Children students in selected schools
* Anthropometric diagnostic of normality or overweight
* Informed consent of parents

Exclusion Criteria:

* Children with special diet or children with limited motor functioning

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 0, 12 months
  We will evaluate the change in body mass index

SECONDARY OUTCOMES:
Change in vegetal and fruit consumption | 0, 12 months
  We will evaluate the change in frequency of consumption of diverse fruits and vegetables

OTHER OUTCOMES:
Adiposity | 0, 12 months
  We will evaluate the change in percent of fat mass
Physical activity | 0, 12 months
  We will evaluate the change in the frequency and kinf of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Marco A González, Master, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico